CLINICAL TRIAL: NCT00284830
Title: Search AV Extension and Managed Ventricular Pacing for Promoting Atrio-Ventricular Conduction (SAVE PACe)
Brief Title: SAVEPACe - Search AV Extension and Managed Ventricular Pacing for Promoting Atrio-Ventricular Conduction
Acronym: SAVEPACe
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Cardiac Rhythm and Heart Failure (Industry)
Responsible Party: Medtronic CRDM Clinical Research, Medtronic CRDM Clinical Research
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 191
Record Dates: First submitted 2006-01-31; First posted 2006-02-01 (Estimated); Last update posted 2008-02-29 (Estimated); Status verified 2008-02

CONDITIONS: Sick Sinus Syndrome; Heart Failure, Congestive; Atrial Fibrillation; Bradycardia; Ventricular Dysfunction
Keywords: Right Ventricular Pacing; Persistent Atrial Fibrillation; Atrioventricular Conduction; Heart Failure Hospitalization; Cardiovascular Health Care Utilization; Sinus-node Disease; Minimized Ventricular Pacing
MeSH Terms: conditions — Sick Sinus Syndrome; Heart Failure; Atrial Fibrillation; Bradycardia; Ventricular Dysfunction

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): dual-chamber minimal ventricular pacing with the use of new pacemaker features designed to promote atrioventricular conduction, preserve ventricular conduction, and prevent ventricular desynchronization
  Interventions: Device: Implantable Pulse Generators
- 2 (No Intervention): conventional dual-chamber pacing

INTERVENTIONS:
Device: Implantable Pulse Generators — dual-chamber minimal ventricular pacing with the use of new pacemaker features designed to promote atrioventricular conduction, preserve ventricular conduction, and prevent ventricular desynchronization
  Other Names: Search AV+; Search AV; MVP; Medtronic; Dual-Chamber Pacemaker
  Arms: 1

SUMMARY:
SAVE PACe is a large, prospective, single-blinded, randomized clinical trial with the main objective to study the effect of unnecessary right ventricular apical pacing on the clinical outcome of time to development of persistent AF.

DETAILED DESCRIPTION:
Conventional dual-chamber pacing maintains atrioventricular synchrony but results in high percentages of ventricular pacing, which causes ventricular desynchronization and has been linked to an increased risk of atrial fibrillation in patients with sinus-node disease.

Patients with sinus-node disease and intact atrioventricular conduction are randomly assigned to receive conventional dual-chamber pacing or dual-chamber minimal ventricular pacing with the use of new Medtronic pacemaker features designed to promote atrioventricular conduction, preserve ventricular conduction, and prevent ventricular desynchronization. The primary end point was time to persistent atrial fibrillation.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age and older
* Willing and able to give informed consent
* Willing and able to comply with the study follow-up schedule
* Class I/ClassII indications for dual chamber pacing
* Initial implant of a Kappa 700, Kappa 900, EnPulse, or EnRhythm dual chamber IPG
* Demonstrate 1 to 1 conduction and a QRS interval of < 120ms at 100 beats per minutes for a period of nine seconds while atrial pacing

Exclusion Criteria:

* Less than 18 years of age
* Unwilling or unable to give informed consent
* Unwilling or unable to commit to follow-up schedule
* Medical conditions that would preclude the testing required by the protocol or limit study participation
* Enrolled or intend to participate in another clinical trial during the course of this study
* A life expectancy of less than 2 years
* History of continuous atrial fibrillation for the 6 months prior to screen visit
* Two or more cardioversions, chemical or electrical, within the past 6 months prior to screen
* History of persistent second or third degree atrioventricular block
* A prior implant of pacemaker or defibrillator device
* A baseline, pre-paced QRS >120 ms on surface ECG
* Failure of the 1 to 1 atrioventricular conduction test
* Anticipated major cardiac surgery within the course of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1070 (Actual)
Dates: Start 2003-01; Primary Completion 2006-12 (Actual); Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
To compare the time to development of persistent AF between all randomized subjects in the ON and OFF arms. | from Jan 2003 to Dec 2006

SECONDARY OUTCOMES:
To compare composite endpoint of AF and heart failure hospitalization (HFH), HFH, cardiovascular health care utilization, symptoms, HF medications, cumulative %, adverse events and incidence of stroke between the arms. | from Jan 2003 to Dec 2006

CONTACTS AND LOCATIONS:
Overall Officials: Michael O. Sweeney, MD, Principal Investigator — Brigham and Women's Hospital
Locations (67):
- United States (63):
  - Phoenix, Arizona
  - Scottsdale, Arizona
  - Conway, Arkansas
  - Glendale, California
  - La Mesa, California
  - Santa Rosa, California
  - Boulder, Colorado
  - Denver, Colorado
  - Clearwater, Florida
  - Ft. Pierce, Florida
  - Lakeland, Florida
  - Miami Beach, Florida
  - Orlando, Florida
  - Verro Beach, Florida
  - Atlanta, Georgia
  - Tifton, Georgia
  - Maywood, Illinois
  - Rockford, Illinois
  - Lexington, Kentucky
  - Lacombe, Louisiana
  - Annapolis, Maryland
  - Salisbury, Maryland
  - Boston, Massachusetts
  - Worcester, Massachusetts
  - Ann Arbor, Michigan
  - Grand Rapids, Michigan
  - Saint Joseph, Michigan
  - Southfield, Michigan
  - Minneapolis, Minnesota
  - Saint Cloud, Minnesota
  - Saint Paul, Minnesota
  - Tupelo, Mississippi
  - St Louis, Missouri
  - Hastings, Nebraska
  - Cherry Hill, New Jersey
  - Elmer, New Jersey
  - Albuquerque, New Mexico
  - East Syracuse, New York
  - Johnson City, New York
  - New Hyde Park, New York
  - Syracuse, New York
  - The Bronx, New York
  - Charlotte, North Carolina
  - Durham, North Carolina
  - Gastonia, North Carolina
  - Bismarck, North Dakota
  - Cincinnati, Ohio
  - Kettering, Ohio
  - Mansfield, Ohio
  - Toledo, Ohio
  - Corvallis, Oregon
  - Salem, Oregon
  - Easton, Pennsylvania
  - Philadelphia, Pennsylvania
  - York, Pennsylvania
  - Cookeville, Tennessee
  - Germantown, Tennessee
  - Nashville, Tennessee
  - Austin, Texas
  - Houston, Texas
  - Plano, Texas
  - Tyler, Texas
  - Richmond, Virginia
- Canada (4):
  - Vancouver, British Columbia
  - Winnipeg, Manitoba
  - Sainte-Foy, Quebec
  - Trois-Rivières, Quebec

REFERENCES:
- [Result] Sweeney MO, Bank AJ, Nsah E, Koullick M, Zeng QC, Hettrick D, Sheldon T, Lamas GA; Search AV Extension and Managed Ventricular Pacing for Promoting Atrioventricular Conduction (SAVE PACe) Trial. Minimizing ventricular pacing to reduce atrial fibrillation in sinus-node disease. N Engl J Med. 2007 Sep 6;357(10):1000-8. doi: 10.1056/NEJMoa071880. PMID 17804844